CLINICAL TRIAL: NCT04183842
Title: Evaluation of a Fixed Combination of Herbal Extracts to Prevent Symptoms Alcohol-induced Hangovers : A Randomized, Double Blind Placebo Controlled Crossover Study.
Brief Title: Evaluation of a Fixed Combination of Herbal Extracts to Prevent Symptoms Alcohol-induced Hangovers
Acronym: LACIME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Incara Lab (Industry)
Collaborators: Phytomed AB (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PM-2019-03
Record Dates: First submitted 2019-10-16; First posted 2019-12-03 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: Headache; Nausea; Dizziness; Sleepiness; Anxiety; Thirst
MeSH Terms: conditions — Headache; Nausea; Dizziness; Sleepiness; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Randomized, double blind, placebo controlled, crossover study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization chart Code number for Product / Placebo distribution
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LACIME Anti-hangover (Experimental): Combination of plant extracts under liquid form. Oral administration. Dosage 100 ml. To drink 1h00 before alcohol intake together with meal.
  Interventions: Dietary Supplement: LACIME Anti-hangover
- Placebo (Placebo Comparator): Carrot juice under liquid form. Oral administration. Dosage 100 ml. To drink 1h00 before alcohol intake together with meal.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: LACIME Anti-hangover — LACIME Anti-hangover contains the following excipients:
  * Purified water,
  * Xanthan gum,
  * Glycerin,
  * Potassium sorbate (as a preservative)
  * Citric acid (acidity regulator)
  * Aroma (flavouring agent)
  LACIME Anti-hangover contains the following plant extracts and vitamin:
  * Curcuma longa rhizome extract (Curcuma),
  * Panax quinquefolius extract (Ginseng panax),
  * Malpighia punicifolia extract (Acerola),
  * Silybum marianum extract (Milk thistle),
  * Desmodium adscendens extract (Desmodium),
  * Pyridoxine chlorhydrate (Vitamin B6).
  Arms: LACIME Anti-hangover
Other: Placebo — Placebo contains the following excipients :
  * Purified water,
  * Xanthan gum,
  * Glycerin,
  * Potassium sorbate (as a preservative)
  * Citric acid (acidity regulator)
  * Aroma (flavouring agent)
  Placebo contains :
  - Carrot juice
  Arms: Placebo

SUMMARY:
The primary objective of the study is to test whether the tested Product LACIME Anti-hangover is effective in preventing the signs and symptoms of alcohol-induced hangover (such as headache, impaired memory, depression, anxiety, weakness, trouble sleeping and concentrating, nausea, dizziness, sleepiness, thirsty, dry mouth, sweating, sensitivity to light and sounds, vision problems) in healthy subjects.

DETAILED DESCRIPTION:
LACIME Anti-hangover is a food supplement under the form of a syrup (water/glycerin based) containing plan extracts, each one having choleretic properties.

40 healthy subjects will be tested in a randomized, double-blind, placebo-controlled, crossover trial.

The participants will have to attend the 2 phases of the study during which they will receive in a blind way a product (LACIME Anti-hangover or PLACEBO):

If a participant has received LACIME Anti-hangover for Phase 1, the same participant will receive the PLACEBO for Phase 2 and vice versa.

Inclusion Criteria:

For inclusion in the study subjects must fulfil all the following criteria:

20-30 years old healthy males and females, Body weight (kg): 60 - 80 in man and 60-70 in women, People who consume alcohol occasionally and who already have to deal with hangovers Healthy volunteers who consume alcohol regularly and moderately, Having given their free, informed and express consent in writing Co-operative, informed of the need and duration of the controls which make it possible to achieve full adherence to the protocol in place.

Exclusion Criteria:

Excluded from participating in the study:

Volunteers consuming larger amounts of alcohol (more than 2 glasses of alcohol per day) Volunteers taking medication or food supplements that may affect alcohol metabolism.

Women who are pregnant or breastfeeding or plan to become pregnant during the study Subjects with illnesses which may conflict with the investigator's interpretation, if the subject participated in the study Subject planning to change his/her lifestyle during the study (diet, physical activity, etc.) Smoker Subject participating in another study during the clinical study period.

* At the first medical visit all volunteers will be checked for illegibility, randomized, and sign written informed consent including an obligation that they will not take alcohol within the next week and come to the study site a week later at least 3 hours after the last meal.
* At the second visit, participants will attend the study site, where each will fill Hangover Severity Symptoms (HSS) form, donate blood and urine for initial analysis.

Then participants take the Product LACIME Anti-hangover or PLACEBO and after 1hour will start to consume alcohol during two hours with meal (3 sandwiches with cheese or ham) on each of the 2 study phases.

Drink consumption, the composition and sequence:

300 ml of Brandy (41% vol. alcohol) corresponding to an intake of 123 ml or 99 g of alcohol 300 ml of Champagne (13% vol. alcohol) corresponding to an intake of 40 ml or 32 g of alcohol This will ensure a 100% hangover syndrome and a total intake of 131 g of alcohol (a dose of approximately 2 g / kg).

Such a dose will provide a peak concentration after 1 hour and should allow to determine the alcohol 15 hours after absorption.

Smaller doses are usually not detectable after 10-12 hours. (Jones, 2008).

D2 test, blood sampling and urine sampling under medical control is achieved before alcohol intake.

D2 test, blood sampling and urine sampling under medical control is achieved 1h, 4h and 15h after alcohol consumption.

ELIGIBILITY:
Inclusion Criteria:

* 20-30 years old healthy males,
* Body weight (kg): 60 kg - 80 kg in man,
* People who consume alcohol occasionally,
* People who already had to deal with hangovers,
* Healthy volunteers who consume alcohol regularly and moderately,
* Having given their free, informed and express consent in writing,
* Co-operative, informed of the need and duration of the controls which make it possible to achieve full adherence to the protocol in place.

Exclusion Criteria:

* Volunteers consuming larger amounts of alcohol (more than 2 glasses of alcohol per day)
* Volunteers taking medication or food supplements that may affect alcohol metabolism,
* Subjects with illnesses which may conflict with the investigator's interpretation, if the subject participated in the study,
* Subject planning to change his lifestyle during the study (diet, physical activity, etc.)
* Subject participating in another study during the clinical study period.

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-07-04 (Actual); Primary Completion 2019-08-26 (Actual); Study Completion 2019-09-07 (Actual)

PRIMARY OUTCOMES:
Evaluation of the difference in Hangover Severity Scores between the activity of LACIME Anti-hangover and the activity of PLACEBO. | Total duration 2 days (Total=16h00: From 1h00 before alcohol intake until 15h after alcohol consumption)
  Evaluation of the difference in Hangover Severity Scores between the activity of LACIME Anti-hangover and the activity of PLACEBO.
  The measure is the true change in self assessment scores from their baseline. 12 self assessed parameters :
  * Headache,
  * Fatigue, weakness
  * Thirsty
  * Dry mouth
  * Nausea
  * Vomiting
  * Trembling
  * Sweat
  * Depressed
  * Anxiety
  * Trouble Sleeping
  * Sensitivity to light
  For each of the above symptoms, the Hangover Severity Scale ranges from 0 to 4.
  The Scores are evaluated according to the following:
  * Absent=0
  * Mild=1
  * Moderate=2
  * Severe=3
  * Incapacitating=4
  Self assessment is achieved:
  * Day 1 : 1h00 before alcohol intake (baseline)
  * Day 1 : Alcohol and meal intake
  * Day 1 : 1h00 after alcohol intake (Visit 1a)
  * Day 1 : 4h00 after alcohol intake (Visit 1b)
  * Day 1 : 15h00 after alcohol intake (Visit 1c)

SECONDARY OUTCOMES:
Evaluation of the difference in Cognitive Performance Score between the activity of LACIME Anti-hangover and the activity of PLACEBO according to "d2" psychometric test. | Total duration 2 days (Total=16h00: From 1h00 before alcohol intake until 15h after alcohol consumption)
  The test "d2" consists of identifying and marking the letters "d" accompanied by two dashes only in the middle of other annoying characters.
  The test "d2" is an array containing 14 lines of 47 characters which must all be checked.
  The recorded figures are :
  * correctly identifyed characters,
  * omissions,
  * confusions,
  * total number of errors.
  Three indices, reveal the evolution of the concentration:
  * Concentration Performance (error-corrected processing rate)
  * Speed of treatment
  * Fluctuation Rate (precision in treatment and accuracy)
  Changes of psychometric parameters are evaluated by d2 test at:
  * Day 1 : 1h00 before alcohol intake (baseline)
  * Day 1 : Alcohol and meal intake
  * Day 1 : 1h00 after alcohol intake (Visit 1a)
  * Day 1 : 4h00 after alcohol intake (Visit 1b)
  * Day 1 : 15h00 after alcohol intake (Visit 1c)
Acetaldehyde blood assay (Jones, 2008) | Total duration 2 days (Total=16h00: From 1h00 before alcohol intake until 15h after alcohol consumption)
  Alcohol is mainly metabolized by hepatic oxydation by NADH / NAD+ enzymatic route.
  Ingestion of Alcohol provoques an increase in the ratio NADH / NAD+ which disrupts all the other metabolic pathways in equilibrium with this coenzyme.
  In the first stage of hepatic metabolism, the enzyme dehydrogenase converts alcohol into Acetaldehyde, a very toxic substance that has effects on the entire body.
  Acetaldehyde is a choice marker to evaluate the level of alcoholic intoxication whenever it is an acute, massive or chronic absorption.
  Titration of blood concentration of Acetaldehyde in mg/l
  Changes of blood parameters from baseline are evaluated at:
  * Day 1 : 1h00 before alcohol intake (baseline)
  * Day 1 : Alcohol and meal intake
  * Day 1 : 1h00 after alcohol intake (Visit 1a)
  * Day 1 : 4h00 after alcohol intake (Visit 1b)
  * Day 1 : 15h00 after alcohol intake (Visit 1c)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander PANOSSIAN, Pr., Dr, Study Chair — Swedish Herbal Institute AB; Areg HOVHANNISYAN, PhD, Dr.Sci, Study Director — Head od National Anti-Doping Organization; Artur POTOSSIAN, Dr. MD, Principal Investigator — CARDIOMED Family Health Center; Samvel HAYRUMYAN, PhD, MD, Principal Investigator — CARDIOMED Family Health Center
Locations (1):
- Unimed Medical Center, Abovyan, Yerevan, Armenia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 2 months after study completion for 6 months.
Access Criteria: Data access is controlled by the Central Contact Person. Please contact bommelaer@shadeline.com for Password
URL: https://hidrive.ionos.com/share/bv7z7738u3

REFERENCES:
- [Background] Aziz AM, Brothers S, Sartor G, Holm L, Heilig M, Wahlestedt C, Thorsell A. The nociceptin/orphanin FQ receptor agonist SR-8993 as a candidate therapeutic for alcohol use disorders: validation in rat models. Psychopharmacology (Berl). 2016 Oct;233(19-20):3553-63. doi: 10.1007/s00213-016-4385-8. Epub 2016 Aug 11. PMID 27515665
- [Background] Economidou D, Cippitelli A, Stopponi S, Braconi S, Clementi S, Ubaldi M, Martin-Fardon R, Weiss F, Massi M, Ciccocioppo R. Activation of brain NOP receptors attenuates acute and protracted alcohol withdrawal symptoms in the rat. Alcohol Clin Exp Res. 2011 Apr;35(4):747-55. doi: 10.1111/j.1530-0277.2010.01392.x. Epub 2011 Jan 11. PMID 21223310
- [Background] Jayawardena R, Thejani T, Ranasinghe P, Fernando D, Verster JC. Interventions for treatment and/or prevention of alcohol hangover: Systematic review. Hum Psychopharmacol. 2017 Sep;32(5). doi: 10.1002/hup.2600. Epub 2017 May 31. PMID 28568743
- [Background] Kim H, Kim YJ, Jeong HY, Kim JY, Choi EK, Chae SW, Kwon O. A standardized extract of the fruit of Hovenia dulcis alleviated alcohol-induced hangover in healthy subjects with heterozygous ALDH2: A randomized, controlled, crossover trial. J Ethnopharmacol. 2017 Sep 14;209:167-174. doi: 10.1016/j.jep.2017.07.028. Epub 2017 Jul 24. PMID 28750942
- [Background] Lee HS, Isse T, Kawamoto T, Baik HW, Park JY, Yang M. Effect of Korean pear (Pyruspyrifolia cv. Shingo) juice on hangover severity following alcohol consumption. Food Chem Toxicol. 2013 Aug;58:101-6. doi: 10.1016/j.fct.2013.04.007. Epub 2013 Apr 13. PMID 23587660
- [Background] Lee MH, Kwak JH, Jeon G, Lee JW, Seo JH, Lee HS, Lee JH. Red ginseng relieves the effects of alcohol consumption and hangover symptoms in healthy men: a randomized crossover study. Food Funct. 2014 Mar;5(3):528-34. doi: 10.1039/c3fo60481k. PMID 24458173
- [Background] Pittler MH, White AR, Stevinson C, Ernst E. Effectiveness of artichoke extract in preventing alcohol-induced hangovers: a randomized controlled trial. CMAJ. 2003 Dec 9;169(12):1269-73. PMID 14662662
- [Background] Robertson BM, Piasecki TM, Slutske WS, Wood PK, Sher KJ, Shiffman S, Heath AC. Validity of the hangover symptoms scale: evidence from an electronic diary study. Alcohol Clin Exp Res. 2012 Jan;36(1):171-7. doi: 10.1111/j.1530-0277.2011.01592.x. Epub 2011 Jul 18. PMID 21762183
- [Background] Slutske WS, Piasecki TM, Hunt-Carter EE. Development and initial validation of the Hangover Symptoms Scale: prevalence and correlates of Hangover Symptoms in college students. Alcohol Clin Exp Res. 2003 Sep;27(9):1442-50. doi: 10.1097/01.ALC.0000085585.81711.AE. PMID 14506405
- [Background] Wiese J, McPherson S, Odden MC, Shlipak MG. Effect of Opuntia ficus indica on symptoms of the alcohol hangover. Arch Intern Med. 2004 Jun 28;164(12):1334-40. doi: 10.1001/archinte.164.12.1334. PMID 15226168
- Available data/document: Protocol, Validation of Ethic Comitee, Informed consent form, D2 test of attention, Hangover severity scale, Randomization chart — https://hidrive.ionos.com/share/bv7z7738u3 — Password will be provided by Administrator. Please ask for it at : bommelaer@shadeline.com